CLINICAL TRIAL: NCT02254395
Title: PINS Stimulator System for Deep Brain Stimulation to Treat Obesity
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PINS-010
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Brain Stimulation (Experimental): Stimulation is on.
  Interventions: Device: Deep Brain Stimulation
- Placebo (Sham Comparator): Sham Stimulation: Stimulation is off.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation
  Other Names: PINS Stimulator System

SUMMARY:
The purpose of this clinical study is to verify the long term effecacy and safety of a bilateral deep brain stimulation (DBS) produced by Beijing PINS Medical Co., Ltd. as a treatment option for patients with obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18 to 65.
2. Body Mass Index [BMI] >40 kg/m2.

Exclusion Criteria:

1. Medical contraindications for general anesthesia, craniotomy, or DBS surgery
2. Evidence of neurological disorders, e.g., multiple sclerosis, Parkinson's disease and ischemic stroke, or severe brain atrophy or the presence of subdural hygromas or subdural hematomas.
3. Participate in other clinical trial;
4. Has a life expectancy of < 1 year.
5. The investigator and/or enrollment review committee, would preclude participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Body Weight | 12 month
  Body weight will be recorded at every follow-up visit.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 12 month
Food Intake | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Li Luming, PhD, Study Chair — Tsinghua University